CLINICAL TRIAL: NCT00820586
Title: Intramyocardial Delivery of Autologous Bone Marrow
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: No more funding support for additional procedures
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Antonio Colombo, Director of Invasive Cardiology Unit, IRCCS San Raffaele
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TVICPR-003
Record Dates: First submitted 2009-01-08; First posted 2009-01-12 (Estimated); Last update posted 2012-02-02 (Estimated); Status verified 2012-02

CONDITIONS: Refractory Angina
Keywords: Intramyocardial; Autologous; Bone; Marrow; Randomized; Percutaneous; CD34+; Refractory; Angina; Pectoris.
MeSH Terms: conditions — Angina Pectoris

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mononuclear bone marrow derived cells (Experimental): Intramyocardial injection of total mononuclear bone marrow derived cells
  Interventions: Procedure: Mononuclear bone marrow derived cells
- Selected CD34+ bone marrow derived cells (Experimental): Intramyocardial injection of selected CD34+ bone marrow derived cells
  Interventions: Procedure: Mononuclear bone marrow derived cells

INTERVENTIONS:
Procedure: Mononuclear bone marrow derived cells — Direct intramyocardial percutaneous delivery of autologous bone marrow-derived total mononuclear cells or selected CD34+ cells
  Other Names: Selected CD34+ bone marrow derived cells

SUMMARY:
A randomized study to assess the safety, feasibility and effectiveness of direct intramyocardial percutaneous delivery of autologous bone marrow-derived total mononuclear cells or selected CD34+ cells in patients with refractory angina pectoris.

DETAILED DESCRIPTION:
Primary Endpoint: Incidence of major adverse cardiac events (MACE) at 30 days. MACE is defined as a combined endpoint of death, acute MI (Q-wave and non-Q wave), revascularization procedures (percutaneous or surgical), and peri-procedural complications (that is, left ventricular perforation with hemodynamic consequences requiring pericardiocentesis, and stroke).

Incidence of MACE at 3, 6 and 12 months

Secondary Endpoints:

* Change in Canadian Cardiovascular Society (CCS) angina classification score from baseline to 12 months
* Changes in the quality of life, as assessed according to the Seattle Angina Questionnaire
* Change in exercise duration and exercise tolerance using standardized treadmill exercise testing from baseline, to 6 months and to 12 months
* Cumulative number of hospitalizations for coronary ischemia and congestive heart failure at 12 months following treatment.
* SPECT-chances in global and regional radionuclide perfusion at rest, peak stress, and redistribution for baseline to 1, 6 and 12 months
* Change in angiographic collateral score at 6 months
* Change in global and regional myocardial contractility (assessed by echocardiography) at baseline, 6 and 12 months.

ELIGIBILITY:
Inclusion criteria:

1. Subjects >21 years old;
2. Subjects with functional class (CCS) III or IV angina;
3. Subjects with left ventricular (LV) ejection fraction ³ 30%
4. Attempted "best" tolerated medical therapy
5. Clinical signs and symptoms of myocardial ischemia with reversible ischemia on perfusion imaging;
6. Patient deemed to be a poor candidate or at high surgical risk;
7. Subject must be able to complete a minimum of 2 minutes but no more than 10 minutes exercise test (Bruce Protocol);
8. Subject (or their legal guardian) understands the nature of the procedure and provides written consent prior to the procedure;
9. Subject is willing to comply with specified follow-up evaluations;
10. Patient must develop angina and a horizontal or down-sloping ST-segment depression of ³ 1 mm during exercise, compared to pre-exercise ST segment, 80 ms from the J point or moderate angina with or without the above ST segment changes.

Angiographic Inclusion Criteria:

1. Severe obstruction (lumen diameter stenosis > 70%) in a coronary or surgical conduit felt to be solely or partially responsible for angina and myocardial ischemia;
2. There must be at least one coronary or surgical conduit with < 70% diameter stenosis
3. Poor candidate for percutaneous coronary intervention of treatment zone
4. Poor candidates for surgical revascularization procedures, such as inadequate target coronary anatomy or lack of potential surgical conduits.

Exclusion Criteria:

1. Pregnant women;
2. Left ventricular ejection fraction <30% as assessed by either echocardiography or left ventriculography;
3. Severe cardiac heart failure with NYHA functional class III-IV symptoms;
4. Chronic atrial fibrillation;
5. Prosthetic aortic valve;
6. Severe (grade III-IV) mitral or aortic insufficiency;
7. Wall thickness of <8 mm (defined by echocardiography) of the proposed target region of myocardium;
8. Severe co-morbidity associated with a reduction in life expectancy of <1 year, such as chronic medical illnesses
9. Braunwald class II unstable angina
10. Severe peripheral (or aortic) vascular disease which might increase the risk of vascular complications (perforation, dissection or embolization);
11. Significant aortic valve pathologic sclerosis or stenosis
12. LV thrombus (mobile or mural-based) seen on echocardiography;
13. Recent (within 4 weeks) documented myocardial infarction (Q and/or non-Q wave) defined as CK-MB >3times upper normal level;
14. Currently enrolled in another investigational device or drug trial that has not completed the required follow-up period;
15. Thrombocytopenia or history of heparin-induced thrombocytopenia or thrombocytosis
16. Leukopenia
17. Leukocytosis
18. Anemia or erythrocytosis
19. Active peptic ulcer or active gastrointestinal bleeding;
20. Chronic renal failure requiring dialysis;
21. Prior or current malignancy
22. Other conditions that can significantly affect the bone-marrow
23. Evidence of concurrent infection (WBC >12.000 mm3, temperature >38.5° C);
24. Serological of clinical evidence of HIV
25. Immunotherapy
26. Abnormal bone-marrow morphology as evident in bone-marrow smear prior to the intervention

Angiographic/Ventriculographic Exclusion Criteria:

1. LV thrombus (mobile or mural-based) seen on left ventriculography;
2. Coronary lesions suitable for percutaneous coronary interventions;
3. Unprotected left main coronary artery disease

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2007-05; Primary Completion 2011-01 (Actual); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of major adverse cardiac events (MACE), defined as a combined endpoint of death, acute MI (Q-wave and non-Q wave), revascularization procedures and peri-procedural complications. | 1, 6, 12 months

SECONDARY OUTCOMES:
Change in Canadian Cardiovascular Society (CCS) angina classification score | 12 months
Changes in the quality of life, as assessed according to the Seattle Angina Questionnaire | 1,3,6,12 months and every year for 8 years
Change in exercise duration and exercise tolerance using standardized treadmill exercise testing | 6,12 months
Cumulative number of hospitalizations for coronary ischemia and congestive heart failure | 12 months
SPECT-chances in global and regional radionuclide perfusion at rest, peak stress, and redistribution | 1, 6, 12 months
Change in angiographic collateral score | 6 months
Change in global and regional myocardial contractility (assessed by echocardiography) | 6, 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS S. Raffaele, Milan, Italy

REFERENCES:
- [Background] Losordo DW, Vale PR, Isner JM. Gene therapy for myocardial angiogenesis. Am Heart J. 1999 Aug;138(2 Pt 2):S132-41. doi: 10.1016/s0002-8703(99)70333-9. PMID 10426872
- [Background] Simons M, Bonow RO, Chronos NA, Cohen DJ, Giordano FJ, Hammond HK, Laham RJ, Li W, Pike M, Sellke FW, Stegmann TJ, Udelson JE, Rosengart TK. Clinical trials in coronary angiogenesis: issues, problems, consensus: An expert panel summary. Circulation. 2000 Sep 12;102(11):E73-86. doi: 10.1161/01.cir.102.11.e73. PMID 10982554
- [Background] Nabel EG, Plautz G, Nabel GJ. Site-specific gene expression in vivo by direct gene transfer into the arterial wall. Science. 1990 Sep 14;249(4974):1285-8. doi: 10.1126/science.2119055.
- [Background] Schumacher B, Pecher P, von Specht BU, Stegmann T. Induction of neoangiogenesis in ischemic myocardium by human growth factors: first clinical results of a new treatment of coronary heart disease. Circulation. 1998 Feb 24;97(7):645-50. doi: 10.1161/01.cir.97.7.645. PMID 9495299
- [Background] Isner JM, Pieczek A, Schainfeld R, Blair R, Haley L, Asahara T, Rosenfield K, Razvi S, Walsh K, Symes JF. Clinical evidence of angiogenesis after arterial gene transfer of phVEGF165 in patient with ischaemic limb. Lancet. 1996 Aug 10;348(9024):370-4. doi: 10.1016/s0140-6736(96)03361-2. PMID 8709735
- [Background] Rosengart TK, Lee LY, Patel SR, Sanborn TA, Parikh M, Bergman GW, Hachamovitch R, Szulc M, Kligfield PD, Okin PM, Hahn RT, Devereux RB, Post MR, Hackett NR, Foster T, Grasso TM, Lesser ML, Isom OW, Crystal RG. Angiogenesis gene therapy: phase I assessment of direct intramyocardial administration of an adenovirus vector expressing VEGF121 cDNA to individuals with clinically significant severe coronary artery disease. Circulation. 1999 Aug 3;100(5):468-74. doi: 10.1161/01.cir.100.5.468. PMID 10430759
- [Background] Vale PR, Losordo DW, Milliken CE, McDonald MC, Gravelin LM, Curry CM, Esakof DD, Maysky M, Symes JF, Isner JM. Randomized, single-blind, placebo-controlled pilot study of catheter-based myocardial gene transfer for therapeutic angiogenesis using left ventricular electromechanical mapping in patients with chronic myocardial ischemia. Circulation. 2001 May 1;103(17):2138-43. doi: 10.1161/01.cir.103.17.2138. PMID 11331253
- [Background] Asahara T, Masuda H, Takahashi T, Kalka C, Pastore C, Silver M, Kearne M, Magner M, Isner JM. Bone marrow origin of endothelial progenitor cells responsible for postnatal vasculogenesis in physiological and pathological neovascularization. Circ Res. 1999 Aug 6;85(3):221-8. doi: 10.1161/01.res.85.3.221. PMID 10436164
- [Background] Kobayashi T, Hamano K, Li TS, Katoh T, Kobayashi S, Matsuzaki M, Esato K. Enhancement of angiogenesis by the implantation of self bone marrow cells in a rat ischemic heart model. J Surg Res. 2000 Apr;89(2):189-95. doi: 10.1006/jsre.2000.5828. PMID 10729249
- [Background] Tomita S, Mickle DA, Weisel RD, Jia ZQ, Tumiati LC, Allidina Y, Liu P, Li RK. Improved heart function with myogenesis and angiogenesis after autologous porcine bone marrow stromal cell transplantation. J Thorac Cardiovasc Surg. 2002 Jun;123(6):1132-40. doi: 10.1067/mtc.2002.120716. PMID 12063460
- [Background] Shintani S, Murohara T, Ikeda H, Ueno T, Sasaki K, Duan J, Imaizumi T. Augmentation of postnatal neovascularization with autologous bone marrow transplantation. Circulation. 2001 Feb 13;103(6):897-903. doi: 10.1161/01.cir.103.6.897. PMID 11171801
- [Background] Fuchs S, Baffour R, Zhou YF, Shou M, Pierre A, Tio FO, Weissman NJ, Leon MB, Epstein SE, Kornowski R. Transendocardial delivery of autologous bone marrow enhances collateral perfusion and regional function in pigs with chronic experimental myocardial ischemia. J Am Coll Cardiol. 2001 May;37(6):1726-32. doi: 10.1016/s0735-1097(01)01200-1. PMID 11345391
- [Background] Tse HF, Kwong YL, Chan JK, Lo G, Ho CL, Lau CP. Angiogenesis in ischaemic myocardium by intramyocardial autologous bone marrow mononuclear cell implantation. Lancet. 2003 Jan 4;361(9351):47-9. doi: 10.1016/S0140-6736(03)12111-3. PMID 12517468
- [Background] Orlic D, Kajstura J, Chimenti S, Jakoniuk I, Anderson SM, Li B, Pickel J, McKay R, Nadal-Ginard B, Bodine DM, Leri A, Anversa P. Bone marrow cells regenerate infarcted myocardium. Nature. 2001 Apr 5;410(6829):701-5. doi: 10.1038/35070587. PMID 11287958
- [Background] Kamihata H, Matsubara H, Nishiue T, Fujiyama S, Amano K, Iba O, Imada T, Iwasaka T. Improvement of collateral perfusion and regional function by implantation of peripheral blood mononuclear cells into ischemic hibernating myocardium. Arterioscler Thromb Vasc Biol. 2002 Nov 1;22(11):1804-10. doi: 10.1161/01.atv.0000039168.95670.b9. PMID 12426208
- [Background] Kawamoto A, Tkebuchava T, Yamaguchi J, Nishimura H, Yoon YS, Milliken C, Uchida S, Masuo O, Iwaguro H, Ma H, Hanley A, Silver M, Kearney M, Losordo DW, Isner JM, Asahara T. Intramyocardial transplantation of autologous endothelial progenitor cells for therapeutic neovascularization of myocardial ischemia. Circulation. 2003 Jan 28;107(3):461-8. doi: 10.1161/01.cir.0000046450.89986.50. PMID 12551872
- [Background] Tateishi-Yuyama E, Matsubara H, Murohara T, Ikeda U, Shintani S, Masaki H, Amano K, Kishimoto Y, Yoshimoto K, Akashi H, Shimada K, Iwasaka T, Imaizumi T; Therapeutic Angiogenesis using Cell Transplantation (TACT) Study Investigators. Therapeutic angiogenesis for patients with limb ischaemia by autologous transplantation of bone-marrow cells: a pilot study and a randomised controlled trial. Lancet. 2002 Aug 10;360(9331):427-35. doi: 10.1016/S0140-6736(02)09670-8. PMID 12241713
- [Background] Assmus B, Schachinger V, Teupe C, Britten M, Lehmann R, Dobert N, Grunwald F, Aicher A, Urbich C, Martin H, Hoelzer D, Dimmeler S, Zeiher AM. Transplantation of Progenitor Cells and Regeneration Enhancement in Acute Myocardial Infarction (TOPCARE-AMI). Circulation. 2002 Dec 10;106(24):3009-17. doi: 10.1161/01.cir.0000043246.74879.cd. PMID 12473544
- [Background] Strauer BE, Brehm M, Zeus T, Kostering M, Hernandez A, Sorg RV, Kogler G, Wernet P. Repair of infarcted myocardium by autologous intracoronary mononuclear bone marrow cell transplantation in humans. Circulation. 2002 Oct 8;106(15):1913-8. doi: 10.1161/01.cir.0000034046.87607.1c. PMID 12370212
- [Background] Perin EC, Dohmann HF, Borojevic R, Silva SA, Sousa AL, Mesquita CT, Rossi MI, Carvalho AC, Dutra HS, Dohmann HJ, Silva GV, Belem L, Vivacqua R, Rangel FO, Esporcatte R, Geng YJ, Vaughn WK, Assad JA, Mesquita ET, Willerson JT. Transendocardial, autologous bone marrow cell transplantation for severe, chronic ischemic heart failure. Circulation. 2003 May 13;107(18):2294-302. doi: 10.1161/01.CIR.0000070596.30552.8B. Epub 2003 Apr 21. PMID 12707230
- [Background] Fuchs S, Satler LF, Kornowski R, Okubagzi P, Weisz G, Baffour R, Waksman R, Weissman NJ, Cerqueira M, Leon MB, Epstein SE. Catheter-based autologous bone marrow myocardial injection in no-option patients with advanced coronary artery disease: a feasibility study. J Am Coll Cardiol. 2003 May 21;41(10):1721-4. doi: 10.1016/s0735-1097(03)00328-0. PMID 12767654
- [Background] Schachinger V, Erbs S, Elsasser A, Haberbosch W, Hambrecht R, Holschermann H, Yu J, Corti R, Mathey DG, Hamm CW, Suselbeck T, Werner N, Haase J, Neuzner J, Germing A, Mark B, Assmus B, Tonn T, Dimmeler S, Zeiher AM; REPAIR-AMI Investigators. Improved clinical outcome after intracoronary administration of bone-marrow-derived progenitor cells in acute myocardial infarction: final 1-year results of the REPAIR-AMI trial. Eur Heart J. 2006 Dec;27(23):2775-83. doi: 10.1093/eurheartj/ehl388. Epub 2006 Nov 10. PMID 17098754
- [Background] Lunde K, Solheim S, Aakhus S, Arnesen H, Abdelnoor M, Egeland T, Endresen K, Ilebekk A, Mangschau A, Fjeld JG, Smith HJ, Taraldsrud E, Grogaard HK, Bjornerheim R, Brekke M, Muller C, Hopp E, Ragnarsson A, Brinchmann JE, Forfang K. Intracoronary injection of mononuclear bone marrow cells in acute myocardial infarction. N Engl J Med. 2006 Sep 21;355(12):1199-209. doi: 10.1056/NEJMoa055706. PMID 16990383
- [Background] Meyer GP, Wollert KC, Lotz J, Steffens J, Lippolt P, Fichtner S, Hecker H, Schaefer A, Arseniev L, Hertenstein B, Ganser A, Drexler H. Intracoronary bone marrow cell transfer after myocardial infarction: eighteen months' follow-up data from the randomized, controlled BOOST (BOne marrOw transfer to enhance ST-elevation infarct regeneration) trial. Circulation. 2006 Mar 14;113(10):1287-94. doi: 10.1161/CIRCULATIONAHA.105.575118. Epub 2006 Mar 6. PMID 16520413
- [Background] Kim MC, Kini A, Sharma SK. Refractory angina pectoris: mechanism and therapeutic options. J Am Coll Cardiol. 2002 Mar 20;39(6):923-34. doi: 10.1016/s0735-1097(02)01716-3. PMID 11897431
- [Background] Mannheimer C, Camici P, Chester MR, Collins A, DeJongste M, Eliasson T, Follath F, Hellemans I, Herlitz J, Luscher T, Pasic M, Thelle D. The problem of chronic refractory angina; report from the ESC Joint Study Group on the Treatment of Refractory Angina. Eur Heart J. 2002 Mar;23(5):355-70. doi: 10.1053/euhj.2001.2706. No abstract available. PMID 11846493
- [Background] Mukherjee D, Bhatt DL, Roe MT, Patel V, Ellis SG. Direct myocardial revascularization and angiogenesis--how many patients might be eligible? Am J Cardiol. 1999 Sep 1;84(5):598-600, A8. doi: 10.1016/s0002-9149(99)00387-2. PMID 10482164
- [Background] Spertus JA, Winder JA, Dewhurst TA, Deyo RA, Prodzinski J, McDonell M, Fihn SD. Development and evaluation of the Seattle Angina Questionnaire: a new functional status measure for coronary artery disease. J Am Coll Cardiol. 1995 Feb;25(2):333-41. doi: 10.1016/0735-1097(94)00397-9. PMID 7829785
- [Background] Vale PR, Losordo DW, Tkebuchava T, Chen D, Milliken CE, Isner JM. Catheter-based myocardial gene transfer utilizing nonfluoroscopic electromechanical left ventricular mapping. J Am Coll Cardiol. 1999 Jul;34(1):246-54. doi: 10.1016/s0735-1097(99)00143-6. PMID 10400018
- [Background] Ben-Haim SA, Osadchy D, Schuster I, Gepstein L, Hayam G, Josephson ME. Nonfluoroscopic, in vivo navigation and mapping technology. Nat Med. 1996 Dec;2(12):1393-5. doi: 10.1038/nm1296-1393. No abstract available. PMID 8946843
- [Background] Kornowski R, Hong MK, Gepstein L, Goldstein S, Ellahham S, Ben-Haim SA, Leon MB. Preliminary animal and clinical experiences using an electromechanical endocardial mapping procedure to distinguish infarcted from healthy myocardium. Circulation. 1998 Sep 15;98(11):1116-24. doi: 10.1161/01.cir.98.11.1116. PMID 9736599
- [Background] Gepstein L, Goldin A, Lessick J, Hayam G, Shpun S, Schwartz Y, Hakim G, Shofty R, Turgeman A, Kirshenbaum D, Ben-Haim SA. Electromechanical characterization of chronic myocardial infarction in the canine coronary occlusion model. Circulation. 1998 Nov 10;98(19):2055-64. doi: 10.1161/01.cir.98.19.2055. PMID 9808605
- [Background] Kornowski R, Hong MK, Leon MB. Comparison between left ventricular electromechanical mapping and radionuclide perfusion imaging for detection of myocardial viability. Circulation. 1998 Nov 3;98(18):1837-41. doi: 10.1161/01.cir.98.18.1837. PMID 9799201
- [Background] Hamano K, Nishida M, Hirata K, Mikamo A, Li TS, Harada M, Miura T, Matsuzaki M, Esato K. Local implantation of autologous bone marrow cells for therapeutic angiogenesis in patients with ischemic heart disease: clinical trial and preliminary results. Jpn Circ J. 2001 Sep;65(9):845-7. doi: 10.1253/jcj.65.845. PMID 11548889
- [Result] Assmus B, Honold J, Schachinger V, Britten MB, Fischer-Rasokat U, Lehmann R, Teupe C, Pistorius K, Martin H, Abolmaali ND, Tonn T, Dimmeler S, Zeiher AM. Transcoronary transplantation of progenitor cells after myocardial infarction. N Engl J Med. 2006 Sep 21;355(12):1222-32. doi: 10.1056/NEJMoa051779. PMID 16990385